CLINICAL TRIAL: NCT02372149
Title: Treatment With Gamunex 10% Intravenous Immunoglobulin (IVIg) for Patients With Demyelination and Diabetes Mellitus: A Blinded, Placebo-Controlled Crossover Pilot Study
Brief Title: IVIg for Demyelination in Diabetes Mellitus
Acronym: IDIDM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Ari Breiner, MD, Assistant Professor of Medicine (Neurology), University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-8297-B
Record Dates: First submitted 2015-02-12; First posted 2015-02-26 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Peripheral Neuropathy; Diabetes Mellitus; Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Diabetes Mellitus; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins, Intravenous; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVIg--Washout--0.9% NaCl (CROSSOVER) (Experimental): 1. 10% caprylate-chromatography purified intravenous immunoglobulin (IVIg) Initial dose: 1.0gm/kg/day for 2 days (maximum 80gm/day). Maintenance dose (monthly x3): 1.0mg/kg/day for 1 day (maximum 80gm/day)
  2. Washout period
  3. 0.9% sodium chloride in water - equal volume to IVIg - Monthly x4
  Interventions: Drug: 10% intravenous immunoglobulin (IVIg); Drug: 0.9% sodium chloride
- 0.9% NaCl--Washout--IVIg (CROSSOVER) (Experimental): 1. 0.9% sodium chloride in water - equal volume to IVIg - Monthly x4
  2. Washout period
  3. 10% caprylate-chromatography purified intravenous immunoglobulin (IVIg) Initial dose: 1.0gm/kg/day for 2 days (maximum 80gm/day). Maintenance dose (monthly x3): 1.0mg/kg/day for 1 day (maximum 80gm/day)
  Interventions: Drug: 10% intravenous immunoglobulin (IVIg); Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: 10% intravenous immunoglobulin (IVIg)
  Other Names: Gamunex
Drug: 0.9% sodium chloride
  Other Names: Normal Saline

SUMMARY:
The purpose of this study is to determine whether intravenous immunoglobulin (IVIg) is an effective intervention for patients with diabetes, peripheral neuropathy, and demyelination on nerve conduction studies. All patients will receive both IVIg and placebo for 3 months each, with a 3 month washout period in between.

DETAILED DESCRIPTION:
There is a knowledge gap with regards to the appropriate method of detecting and treating chronic inflammatory demyelinating polyneuropathy (CIDP), in patients with co-existent diabetes. In this pilot study the investigators plan to examine the overlap between diabetic polyneuropathy and CIDP by treating patients with diabetes and demyelinating abnormalities using IVIg. The investigators will enroll diabetes patients with a broad spectrum of demyelinating abnormalities.

The proposed trial will be an explanatory, blinded, single-centre, superiority, randomized controlled cross-over trial. Each patient will receive 3 months of 10% intravenous immunoglobulin and 3 months of placebo (0.9% sodium chloride in water) with a 3-month washout period. The primary outcome measure is the mean change in ONLS (Overall Neuropathy Limitation Scale), a measure of disability in polyneuropathy; however secondary outcome measures will consider impairments and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Diabetes, as per American Diabetes Association Criteria.
3. Clinical evidence of polyneuropathy and NCS shows 2 separate motor nerves (median, ulnar, tibial, or peroneal) which meet criteria for demyelination, defined as follows:

   1. Conduction velocity <90% lower limit of normal (LLN), distal latency >110% upper limit of normal (ULN), or minimal F-wave latency >110% ULN
   2. The changes are not exclusively due to median neuropathy at the wrist, ulnar neuropathy at the elbow, or peroneal neuropathy at the fibular head.
4. Clinical suspicion of possible demyelinating polyneuropathy (CIDP).

Exclusion Criteria:

1. Pregnant patients, or those of childbearing potential not using contraception.
2. Patients <18 years of age.
3. Presence of an alternative etiology of peripheral neuropathy, such as: hereditary neuropathies (Charcot Marie-Tooth disease); B-vitamin deficiency- or excess-related neuropathy; uremic neuropathy; neuropathy secondary to monoclonal gammopathy; history of cancer- or chemotherapy-related neuropathy; other toxin exposures; and alcoholic neuropathy.
4. Contraindication to IVIg, including: history of recurrent thrombosis, immunoglobulin A deficiency, or severe hypersensitivity reaction to IVIg in past, renal failure, recurrent deep venous thrombosis, pulmonary embolus, stroke, or myocardial infarction.
5. Presence of serious or unstable medical condition, which may preclude study completion or lead to inability to tolerate IVIg. This may include active heart failure, uncontrolled hypertension, or severe anemia, among other conditions.
6. Presence of concomitant neurological illness, which may confound evaluation.
7. Fails or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Change in Overall Neuropathy Limitations Score (ONLS) after 3 months | Baseline and 3 months
  ONLS score will be measured before and after 3 months of IVIg / placebo

SECONDARY OUTCOMES:
Change in Rasch-Built Overall Disability Scale (R-ODS) after 3 months | Baseline and 3 months
  R-ODS score will be measured before and after 3 months of IVIg / placebo
Change in Nerve Conduction Studies (NCS) after 3 months | Baseline and 3 months
  Changes in NCS parameters will be compared before and after 3 months of IVIg / placebo
Change in Medical Research Council (MRC) Sum Score after 3 months | Baseline and 3 months
  MRC sum score will be compared before and after 3 months of IVIg / placebo
Change in Grip Strength after 3 months | Baseline and 3 months
  Grip strength (using Martin vigorimeter) will be compared before and after 3 months of IVIg / placebo
Change in Short Form 36 (SF-36) Quality of Life after 3 months | Baseline and 3 months
  SF-36 will be compared before and after 3 months of IVIg / placebo
Adverse Events | 30 days
  Number of adverse events and serious adverse events within 30 days of IVIg administration

CONTACTS AND LOCATIONS:
Overall Officials: Ari Breiner, MD, FRCPC, Principal Investigator — University of Toronto
Locations (1):
- Toronto General Hospital / Toronto Western Hospital, Toronto, Ontario, Canada